CLINICAL TRIAL: NCT00342446
Title: Follow-Up Study of Women Evaluated and Treated for Infertility
Brief Title: A Follow-up Study of Women Evaluated and Treated for Infertility
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999996019; OH96-C-N019
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2024-01-11 (Actual); Status verified 2024-01

CONDITIONS: Ovarian Cancer; Breast Cancer; Endometrial Cancer; Thyroid Cancer; Colorectal Cancer, Melanoma
Keywords: Gonadotropins; CLOMIPHENE; Ovulation-Stimulating Drugs; Natural History
MeSH Terms: conditions — Ovarian Neoplasms; Breast Neoplasms; Endometrial Neoplasms; Thyroid Neoplasms; Colorectal Neoplasms; Melanoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with Infertility: Patients of all races with primary or secondary infertility, including women with recurrent miscarriages.

SUMMARY:
To assess the relations of infertility causes and treatment to cancer risk, we will conduct a retrospective cohort study of approximately 12,000 women evaluated for infertility between 1965-1988. These women will be ascertained from several large infertility clinics and private practices in various geographic locations in the United States: Boston, Chicago, Detroit, New York, and Palo Alto. These practices were selected on the basis of their having large number of patients who received ovulation stimulating drugs many years in the distant past. Abstractors reviewed clinic medical records to identify eligible study participants and abstract data needed to classify causes of infertility and document therapies employed. Using a variety of tracing sources (including the National Death Index, credit bureaus, and postmasters), the vital status and location of the study subjects were determined. Subjects who were traced and identified as alive are being sent a detailed questionnaire that requests information on their health status as well as on a number of lifestyle practices. For subjects who report a cancer, medical verification is being sought from the diagnosing physicians and/or facilities. Death certificates are being sought for deceased subjects.

DETAILED DESCRIPTION:
BACKGROUND: We previously conducted a retrospective cohort study of 12,193 patients evaluated for infertility between 1960-1988 at five clinical sites. Detailed information abstracted from the medical records, along with questionnaires administered to located patients and cancer incidence and mortality data derived from cancer registries and the National Death Index, allowed us to examine cancer risk related to different causes of infertility and treatments while controlling for other patient characteristics. Although there were some increases of certain cancers related to various causes of infertility, we generally did not observe substantial relationships related to use of different fertility drugs. The one exception was some increased risk of uterine cancers with clomiphene use, of interest given the drug's chemical similarity to tamoxifen. Our numbers of patients with certain cancers (e.g., ovarian, uterine) were, however, limited and we had insufficient power to evaluate subgroup effects (e.g., drug relationships among nulligravid women).

OBJECTIVES: We therefore conducted an updated follow-up of these patients in order to assess cancer risk in relation to causes of infertility and therapeutic regimens used to treat these causes.

ELIGIBILITY: This study gained an additional 10 years of follow-up among the patients deemed eligible for the previous investigation. This included women with both primary and second infertility. Approximately 39% of the cohort previously were prescribed clomiphene citrate, while 10% received gonadotrophins.

DESIGN: Passive follow-up was attempted for patients who previously did not participate and for whom only information available in clinic records could be retained. All other patients were traced for active as well as passive follow-up. Active follow-up involved requesting that patients complete a short questionnaire, whereas passive follow-up was via linkage to cancer registries and the National Death Index. While cancer risks were assessed in relation to the general population, the majority of comparisons were internal ones, involving the calculation of relative risks (RRs) associated with different causes of infertility or treatment regimens while controlling for other cancer risk predictors.

ELIGIBILITY:
* INCLUSION CRITERIA:

The following criteria for inclusion in the study cohort will apply:

Patient is female.

Patient was evaluated for infertility between (and including) 1965 and 1988.

Patient had a U.S. address at the time of evaluation for infertility.

Patient was seen twice by the physician, or was seen once but had a referral from another physician.

Patient's infertility was not due to gonadal dysgenesis or congenital abnormalities of the reproductive system.

Patient's visit to the infertility specialist was not to have a tubal ligation reversed.

Ages: 44 Years to 88 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects were enrolled based on treatment at fertility clinic.@@@
Sampling Method: Non-Probability Sample
Enrollment: 12193 (Actual)
Dates: Start 1995-10-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2023-01-11 (Actual)

PRIMARY OUTCOMES:
Cancer | ongoing
  Breast, endometrial, ovarian, thyroid, melanoma

SECONDARY OUTCOMES:
Mortality | Ongoing
  All cause and cancer-specific death

CONTACTS AND LOCATIONS:
Overall Officials: Gretchen Benson, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- Columbia University, New York, New York, United States

REFERENCES:
- [Background] Bamford PN, Steele SJ. Uterine and ovarian carcinoma in a patient receiving gonadotrophin therapy. Case report. Br J Obstet Gynaecol. 1982 Nov;89(11):962-4. doi: 10.1111/j.1471-0528.1982.tb05067.x. No abstract available. PMID 7171506
- [Background] Carter ME, Joyce DN. Ovarian carcinoma in a patient hyperstimulated by gonadotropin therapy for in vitro fertilization: a case report. J In Vitro Fert Embryo Transf. 1987 Apr;4(2):126-8. doi: 10.1007/BF01555453. No abstract available. PMID 3110335
- [Background] Atlas M, Menczer J. Massive hyperstimulation and borderline carcinoma of the ovary. A possible association. Acta Obstet Gynecol Scand. 1982;61(3):261-3. doi: 10.3109/00016348209156568. PMID 7124357